CLINICAL TRIAL: NCT02727738
Title: Randomized Open Clinical Study to Evaluate the Efficacy of Selenium Plus Methimazole for Treatment of Graves' Hyperthyroidism
Brief Title: Treatment of Graves' Hyperthyroidism With Selenium Plus Methimazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, MD, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPisa
Record Dates: First submitted 2015-06-30; First posted 2016-04-05 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Graves' Disease
Keywords: Hyperthyroidism; Methimazole; Selenium
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Selenium; Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methimazole plus selenium (Experimental): Methimazole 5-30 mg daily for 90 days Selenium 80 bid for 90 days
  Interventions: Dietary Supplement: Selenium; Drug: Methimazole
- Methimazole (Active Comparator): Methimazole 5-30 mg daily for 90 days
  Interventions: Drug: Methimazole

INTERVENTIONS:
Dietary Supplement: Selenium — Selenium 80 mg bid for 90 days
  Other Names: Syrel
  Arms: Methimazole plus selenium
Drug: Methimazole — Methimazole starting dose depending on FT3 values (15 mg/day or 20 mg/day or 30 mg/day, for FT3 values <10 pg/ml, 10-15 pg/ml, >15 pg/ml, respectively) to be tapered by 5 mg/day every 15 days down to values sufficient for FT3 to be normal
  Other Names: Tapazole

SUMMARY:
Evaluation of the efficacy of the combined treatment (methimazole plus selenium) in the control of hyperthyroidism as compared to methimazole alone in 30 Graves' disease (GD) untreated patients.

DETAILED DESCRIPTION:
30 untreated GD hyperthyroid patients will be randomized into two groups (A and B). Group A patients will be treated with an anti-thyroid drug (methimazole) at the dose aimed to control hyperthyroidism. Group B patients will be treated with methimazole plus selenium (160 mg daily). Patients will be evaluated at time 0, 45 and 90 days for symptoms of hyperthyroidism (by a specific questionnaire), clinical status (weight, heart rate), laboratory (thyroid function tests, TSHR autoantibodies, serum selenium, index of oxidative stress-MDA, cholesterol, SHBG) and EKG. The aim of the study is to evaluate if the combined treatment (methimazole plus selenium) is more effective than methimazole alone in controlling GD hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroid untreated Graves' disease patients

Exclusion Criteria:

* Hyperthyroid treated Graves' disease patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Control of hyperthyroidism | 90 days
  Comparison of FT3 and FT4 values (pg/ml) between groups
Clinical manifestations of hyperthyroidism-1 | 90 days
  Comparison of heart rate between groups
Clinical manifestations of hyperthyroidism-2 | 90 days
  Comparison of BMI between groups
Clinical manifestations of hyperthyroidism-3 | 90 days
  Comparison of total serum cholesterol between groups
Clinical manifestations of hyperthyroidism-4 | 90 days
  Comparison of total serum sex hormone binding globulin between groups
Clinical manifestations of hyperthyroidism-5 | 90 days
  Comparison of subjective hyperthyroidism symptoms score collected by questionnaire between groups

SECONDARY OUTCOMES:
Control of hyperthyroidism | 45 days
  Comparison of FT3 and FT4 values (pg/ml) between groups
Clinical manifestations of hyperthyroidism-1 | 45 days
  Comparison of heart rate between groups
Selenium levels | 45 days
  Comparison of serum selenium levels between groups
Selenium levels | 90 days
  Comparison of serum selenium levels between groups
Oxidative stress parameters-1 | 45 days
  Comparison of serum malondialdehyde levels between groups
Oxidative stress parameters-2 | 45 days
  Comparison of serum glutathione peroxidase levels between groups
Thyroid autoimmunity-1 | 45 days
  Comparison of serum anti-thyroperoxidase antibodies levels and prevalence between groups
Thyroid autoimmunity-2 | 45 days
  Comparison of serum anti-thyrotropin receptor antibodies levels and prevalence between groups
Oxidative stress parameters-1 | 90 days
  Comparison of serum malondialdehyde levels between groups
Oxidative stress parameters-2 | 90 days
  Comparison of serum glutathione peroxidase levels between groups
Thyroid autoimmunity-1 | 90 days
  Comparison of serum anti-thyroperoxidase antibodies levels and prevalence between groups
Thyroid autoimmunity | 90 days
  Comparison of serum anti-thyrotropin receptor antibodies levels and prevalence between groups
Adverse events of selenium | 45 days
Adverse events of selenium | 90 days
Clinical manifestatations of hyperthyroidism-2 | 45 days
  Comparison of BMI between groups
Clinical manifestations of hyperthyroidism-3 | 45 days
  Comparison of total serum sex hormone binding globulin between groups
Clinical manifestations of hyperthyroidism-4 | 45 days
  Comparison of subjective hyperthyroidism symptoms score collected by questionnaire between groups

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Marcocci, MD, Principal Investigator — Department of Clinical and Experimental Medicine, University of Pisa
Locations (1):
- Endocrinology Unit, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No